## **Behavioral Activation for Depression: A Randomized Controlled Trial**

Date: November 16<sup>th</sup> 2020

## **Analytic plan**

Mixed Linear Models (MLMs) will account for the hierarchical, dependent nature of the data (repeated measures nested within patients, which again is nested within therapists [if the number of therapists allow for the specification of a level]), testing the time\*group interaction effect, first investigating the effect of treatment compared to the wait-list condition, and then the between-group difference concerning mBA compared to BA. We will also explore the number of recovered patients in BA/mBA vs. waitlist and BA vs mBA according to the minimal clinically important difference for the PHQ-9 (i.e., 5 score points; Lowe, Unutzer, Callahan, Perkins, & Kroenke, 2004) and the reliable change index (Jacobsen & Truax, 1999). In order to determine an effect of treatment through follow-up, groups will be combined and the function of time will be established. The proposed process measures will be explored as mediators of treatment also using MLM evaluated, in separate models, with the products of coefficients method (when comparing groups) and with time-lag analyses (within group). Concerning the experimental data, MLMs will be used to compare the clinical and healthy group from pre to post experimental manipulation at baseline. Comparisons between the clinical group at baseline and the clinical group post-treatment will also be performed, as will an analysis of the within-group effect from pre- to post-treatment among depressed individuals.